CLINICAL TRIAL: NCT03511040
Title: Lumenate Observational Vasospasm Interventional Trial (LOVIT)
Acronym: LOVIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurvana Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR17-006
Record Dates: First submitted 2018-04-10; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Vasospasm, Intracranial; Subarachnoid Hemorrhage
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label, single-arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumenate Intraluminal Device (Experimental): Dilation of vasospastic intracranial vessels
  Interventions: Device: Lumenate Intraluminal Device

INTERVENTIONS:
Device: Lumenate Intraluminal Device — Dilation of vasospastic intracranial vessels
  Other Names: Lumenation

SUMMARY:
The LOVIT study is a European prospective, multi-center, open-label, single-arm feasibility trial designed to determine the safety and angiographic effectiveness through 30 days post treatment with Lumenate Intraluminal Device in the treatment of symptomatic vasospasm.

DETAILED DESCRIPTION:
The Neurvana Lumenate Intraluminal Device is delivered via a percutaneous endovascular approach to the target segment for mechanical assistance and the treatment of vasospasm.

The LOVIT study is a European prospective, multi-center, open-label, single-arm feasibility trial designed to determine the safety and angiographic effectiveness through 30 days post treatment with Lumenate Intraluminal Device in the treatment of symptomatic vasospasm. The primary objective of the study is to support the CE-mark vasospasm label claim for the Lumenate Device. The study will be enrolled at up to 8 European sites with study subjects being followed for 90 days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Subject has the necessary mental capacity to participate and is willing and able to comply with protocol requirements
3. Patient has suffered SAH from a ruptured intracranial aneurysm
4. Has mWFNS ≤3 upon admission to the treating hospital or mWFNS ≤3 after insertion of an endoventricular drain (EVD) for acute hydrocephalus secondary to SAH.
5. Subject has provided written informed consent using the IRB/Ethics committee-approved consent form and are willing to comply with the study protocol and planned follow-ups.
6. Patients that develop symptoms of cerebral vasospasm, as determined by the physician, and/or have diagnostic (e.g. TCD) or radiological evidence of moderate/severe vasospasm.

Exclusion Criteria:

1. Patients that have angiographically confirmed (CTA/MRA) vasospasm at admission to the treating hospital
2. Subjects who require surgical treatment of culprit aneurysm.
3. Endovascular treatment of culprit aneurysm resulting in severe procedural complication (e.g., vessel rupture, embolization or other complication).
4. Placement of intraluminal stent or flow diverter is used to treat culprit aneurysm.
5. Intraluminal stent or flow diverter placed in the 6 months prior to culprit aneurysm rupture.
6. Treated with Intra Arterial vasodilators prior to Lumenate procedure
7. Receiving Anti-coagulant with half-life longer than 24 hours, or Dual antiplatelet therapy (DAPT) including P2Y12 inhibition
8. Woman of child-bearing potential who cannot provide a negative pregnancy test.
9. Patients with vasculitis or connective tissue disorders that put them at risk for vasculitis.
10. Known use of cocaine or methamphetamine within the last month.
11. Any comorbid disease or medical condition with a life expectancy ≤3 months.
12. Known allergy or contraindication to aspirin, heparin, local or general anesthesia
13. Known history of life threatening allergy to contrast dye
14. Serum creatinine ≥2.5 mg/dL
15. Enrollment in another trial involving an investigational product
16. Physician discretion that the patient may not benefit from treatment with Lumenate - reason for exclusion should be documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Vasospasm treatment freedom from complication (Primary Safety Endpoint) | Acute - immediate post-procedure
  No occurrence of device-related procedural complications as assessed by the post treatment angiogram. Catheter angiography will be used to determine the absence/presence of vessel wall disruption (e.g., dissection, perforation) or presence of thrombus within the target vessel.

SECONDARY OUTCOMES:
Vessel caliber change post procedure (Secondary Effectiveness Endpoint) | Acute - immediate post-procedure
  The study's primary effectiveness endpoint is an improvement in the caliber of the treated vasospastic vessel by at least 1 point on the 4-point angiographic scale
Freedom from device-related SAEs at 30 days (Secondary Descriptive Endpoint) | 30±5 days post-procedure
  Any device-related serious adverse events at 30±5 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med Anastasios Mpotsaris, MD, Principal Investigator — Uniklinik RWTH Aachen
Locations (5):
- France (2):
  - Foundation Adolphe de Rothschild, Paris
  - Hospital Purpan, Toulouse
- Uniklinik RWTH Aachen, Aachen, Germany
- National Institute of Neurosciences, Budapest, Hungary
- Karolinska Universitetssjukhuset, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No